CLINICAL TRIAL: NCT06079697
Title: The Effect of Exercise Prehabilitation on Post-Operative Recovery After Head and Neck Cancer Surgery
Brief Title: An Exercise Prehabilitation Intervention for Improving Mobility and Recovery Outcomes in Patients Undergoing Head and Neck Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Ryan Li, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00025357; NCI-2023-07171 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00025357 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2023-09-28; First posted 2023-10-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (prehabilitation) (Experimental): Patients wear a Fitbit or a personal wearable device beginning on day 1 and receive the prehabilitation exercise intervention consisting of 2000-4000 steps per day, sit-to-stand training 3 days per week, and standing therapeutic exercises 3 days per week beginning on day 2 for up to 2-5 weeks prior to surgery. Patients continue wearing the Fitbit or personal wearable device from post-operative day 1 until hospital discharge or until 14 days post-surgery.
  Interventions: Other: Electronic Health Record Review; Other: Exercise Intervention; Other: Medical Device Usage and Evaluation; Other: Survey Administration
- Arm II (usual care) (Active Comparator): Patients wear a Fitbit or personal wearable device beginning on day 1 up until day of surgery and then from post-operative day 1 until hospital discharge or until 14 days post-surgery.
  Interventions: Other: Electronic Health Record Review; Other: Medical Device Usage and Evaluation; Other: Survey Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
Other: Exercise Intervention — Receive prehabilitation exercise intervention
  Arms: Arm I (prehabilitation)
Other: Medical Device Usage and Evaluation — Wear Fitbits
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates a prehabilitation exercise intervention for improving mobility and recovery outcomes in patients undergoing surgery for head and neck cancer. Prehabilitation focuses on optimizing health before surgery in order to improve outcomes after surgery. Prehabilitation may include aspects of nutrition, exercise, mental health, or a combination of these. Exercise has been proven to improve anxiety, depression, fatigue, health related quality of life, and physical function among patients undergoing cancer treatment, as well as cancer survivors. The prehabilitation exercise intervention being studied includes a daily walking program, sit-to-stand training, and standing therapeutic exercises before patients undergo surgery. Receiving this prehabilitation exercise intervention prior to surgery may improve mobility and recovery outcomes in patients after surgery for head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the impact of an exercise prehabilitation program on post-operative outcomes after head and neck cancer surgery.

SECONDARY OBJECTIVE:

I. To evaluate the impact of an exercise prehabilitation program on post-operative weight loss, depression and discharge disposition after head and neck cancer surgery.

EXPLORATORY OBJECTIVES:

I. To evaluate the adherence rate to and satisfaction with a pre-operative exercise prehabilitation program, which will be evaluated at the end of their inpatient stay.

II. To evaluate the impact of lower extremity free tissue transfer on post-operative recovery after undergoing an exercise prehabilitation program, which will be evaluated at the end of their inpatient stay.

III. To evaluate the impact of the duration of prehabilitation on post-operative outcomes after head and neck cancer surgery, which will be evaluated at the end of their inpatient stay.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients wear a Fitbit or personal wearable device beginning on day 1 and receive the prehabilitation exercise intervention consisting of 2000-4000 steps per day, sit-to-stand training 3 days per week, and standing therapeutic exercises 3 days per week beginning on day 2 for up to 2-5 weeks prior to surgery. Patients continue wearing the Fitbit personal wearable device from post-operative day 1 until hospital discharge or until 14 days post-surgery.

ARM II: Patients wear a Fitbit personal wearable device beginning on day 1 up until day of surgery and then from post-operative day 1 until hospital discharge or until 14 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age and younger than 89 years of age. Both men and women and members of all races and ethnic groups may be included
* Planned to undergo major head and neck cancer surgery with free tissue transfer reconstruction at Oregon Health and Science University (OHSU) with the Department of Otolaryngology-Head and Neck Surgery with an expected length of stay (LOS) of 3 days or more
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Non-English speaking
* Planned postoperative admission to the intensive care unit (ICU)
* Social or psychiatric conditions that may interfere with compliance
* Further exclusion criteria may be applied due to conditions that may impact the ability to safely exercise as well as utilize the Fitbit devices:
* Symptoms of or ongoing work-up for unstable angina, uncontrolled tachyarrhythmias, decompensated heart failure, severe aortic stenosis, hypertrophic obstructive cardiomyopathy, uncontrolled hypertension (HTN), uncontrolled pulmonary HTN or uncontrolled asthma
* History of chest pain, dizziness or syncope with exercise
* Bony metastases to the spine or extremities
* Falls in the last year
* Cognitive impairments limiting safety or ability to use technology
* Impaired mobility requiring the use of assistive devices, such as use of a walker or wheelchair at baseline
* Isolation precautions, as they would not be allowed to ambulate on a patient floor post-operatively

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Post-operative mobility | Up to day of discharge or 14 days post-operatively, whichever is sooner.
  Will be measured by daily step counts on the Fitbit or personal wearable device. Descriptive summaries of continuous data will include the sample size, group mean, standard deviation, median, and range. Confidence intervals will be included as appropriate. The primary endpoint of daily post-operative step counts will be compared using two sample t-tests between the intervention and control groups.

SECONDARY OUTCOMES:
Post-operative complications | Up to day of discharge or 14 days post-operatively, whichever is sooner.
  Will be derived from the medical chart, and include pneumonia, DVT, ileus, arrhythmia, wound infection and any events requiring ICU transfer. Descriptive statistics will be used to present the results. A two-sample t-test will be used to analyze continuous variables and Chi-square test will be used for categorical variables.
Length of stay | From post-operative day 1 until day of discharge or 14 days post-operatively, whichever is sooner.
  Derived from the medical record. Descriptive statistics will be used to present the results. A two-sample t-test will be used to analyze continuous variables and Chi-square test will be used for categorical variables.
Depression | Up to day of discharge or 14 days post-operatively, whichever is sooner.
  Measured with the Patient Health Questionnaire-9 (PHQ-9) to determine level of depression on the day of discharge. This screening instrument measures the frequency of 9 signs and symptoms diagnostic of depression, with answers as not at all, several days, more than half of the days, and nearly every day. Total scores range between 0-27, and can indicate mild (<4), moderate (5-14), or severe (>20) depression. Descriptive statistics will be used to present the results. A two-sample t-test will be used to analyze continuous variables and Chi-square test will be used for categorical variables.
Health-related quality of life | Up to day of discharge or 14 days post-operatively, whichever is sooner.
  Measured with the European Organization of Research and Treatment of Cancer Quality of Life Core Questionnaire, version 3.0 (EORTC QLQ C30). A 30-item questionnaire to assess overall quality of life in cancer patients. EORTC QLQ-C30 includes functional scales (physical, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions use 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions use 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged and transformed to 0-100 scale; higher score equates to better level of physical functioning. Descriptive statistics will be used to present the results. A two-sample t-test will be used to analyze continuous variables and Chi-square test will be used for categorical variables.
Weight loss | From time of enrollment to day of discharge or 14 days post-operatively, whichever is sooner.
  Measured in kg. Weight loss will be determined based on their weight at the time of enrollment at initial pre-operative appointment, compared to their weight on the day of discharge. Descriptive statistics will be used to present the results. A two-sample t-test will be used to analyze continuous variables and Chi-square test will be used for categorical variables.
Average daily pain scores | Up to day of discharge or 14 days post-operatively, whichever is sooner.
  Measured on a 1-10 Likert scale, during a patient's inpatient, post-operative stay and obtained from the medical record. Descriptive statistics will be used to present the results. A two-sample t-test will be used to analyze continuous variables and Chi-square test will be used for categorical variables.
Discharge Disposition | At time of discharge or 14 days post-operatively, whichever is sooner.
  Derived from the medical record and may include discharge to home, home with assistance, home with home health, skilled nursing facility, inpatient rehabilitation facility or other facility. Descriptive statistics will be used to present the results. A two-sample t-test will be used to analyze continuous variables and Chi-square test will be used for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Li, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No